CLINICAL TRIAL: NCT02852135
Title: Comparison of LMA Proseal and LMA Supreme for Efficient Ventilation During Lateral Positioned Laparoscopic Surgeries
Brief Title: Comparison of LMA Proseal and LMA Supreme for Efficient Ventilation During Lateral Positioned Laparoscopic Surgeres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Sheng Lan, Principal Investigator, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LMA-lateral-laparoscopic
Record Dates: First submitted 2016-04-16; First posted 2016-08-02 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Urologic Surgical Procedures
Keywords: Laryngeal Mask Airway; lateral position; laparoscopic surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMA Proseal group (Experimental): The patients were randomly allocated to two groups by using computer-generated numbers.In LMA Prosealgroup,LMA Proseal was inserted into each patient after anesthesia induction.
  Interventions: Device: LMA Proseal
- LMA Supreme group (Experimental): The patients were randomly allocated to two groups by using computer-generated numbers.In LMA Supreme group,LMA Supreme was inserted into each patient after anesthesia induction.
  Interventions: Device: LMA Supreme

INTERVENTIONS:
Device: LMA Proseal — After preoxygenation, anaesthesia was induced with propofol, fentanyl and cisatracurium,LMA Proseal was inserted and cuff inflated in each group.
  Arms: LMA Proseal group
Device: LMA Supreme — After preoxygenation, anaesthesia was induced with propofol, fentanyl and cisatracurium ，LMA Supreme was inserted and cuff inflated in each group.
  Arms: LMA Supreme group

SUMMARY:
The LMA Proseal and LMA Supreme are the third generation of LMA with potential advantages over the classic LMA.Several publications have reported the successful, safe use of Laryngeal Mask Airway devices in patients undergoing laparoscopic surgery. However, there have been no studies that have examined the application of LMA in patients during lateral positioned laparoscopic surgery. The aim of this study is to observe the safety and efficacy when LMA Proseal and LMA Supreme used in lateral positioned laparoscopic surgery under general anesthesia.

DETAILED DESCRIPTION:
We undertook a single-blind, parallel-group, randomized controlled trial.The patients were randomized to either LMA Proseal group or LMA Supreme group by computer generated allocation.

The patients were scheduled for elective lateral positioned laparoscopic surgery, such as laparoscopic radical nephrectomy, laparoscopic renal cyst decortication (LRCD) or laparoscopic adrenalectomy.Inclusion criteria for the patients were: Aged>18 years, ASA physical status grade I - Ⅲ and body mass index ≤30 kg.m-2. Exclusion criteria were: anticipated difficult airway (e.g., Modified Mallampati Class IV, oropharyngeal pathology), severe cardiopulmonary disease, increased risk of regurgitation and aspiration (e.g., gastro-esophageal reflux disease, and pregnant patients), and retroperitoneal laparoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* The patients belong to ASA physical status grade I and Ⅲ, aged above 18 years and body weight less than 30 kg/m2,who underwent elective laparoscopic urology surgery in the lateral position.

Exclusion Criteria:

* The patients with anticipated difficult airway (e.g., Modified Mallampati Class IV, oropharyngeal pathology), severe cardiopulmonary disease, increased risk of regurgitation and aspiration (e.g., gastro-esophageal reflux disease, and pregnant patients), and retroperitoneal laparoscopic procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
oropharyngeal seal pressure between LMA Proseal group and LMA Supreme group | intraoperative
  The equilibrating airway pressure was recorded when an audible leak occurred over the mouth.

SECONDARY OUTCOMES:
Ventilatory efficiency scores for the LMAs | intraoperative
Adverse effects in two groups | intraoperative
  The adverse effects including regurgitation,hypoxemia,dysphonia,blood stained after LMA removal, and postoperative sore throat.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Yi, D.M, Study Director — Department of Anesthesiology, Changhai Hospital Shanghai, Shanghai, China, 200433